CLINICAL TRIAL: NCT03880643
Title: Efficacy and Safety of Rituximab in Patients With Refractory Primary Membranous Nephropathy
Brief Title: Rituximab in Refractory Primary Membranous Nephropathy
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Safak Mirioglu, Principal Investigator, Istanbul University
Other Study IDs: 2018/1509
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Glomerulonephritis, Membranous
Keywords: membranous nephropathy; rituximab
MeSH Terms: conditions — Glomerulonephritis, Membranous

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study Group: Patients with primary membranous nephropathy who were treated using rituximab (375 mg/m2/wk for 1-4 weeks) following resistance to at least one set of prior therapies including corticosteroids, alkylating agents or calcineurin inhibitors.

SUMMARY:
Primary membranous nephropathy (PMN), an autoimmune disease mostly associated with anti-phospholipase-A2-receptor (PLA2R) antibodies, is one of the most common causes of nephrotic syndrome in adults. In 30% to 40% of all cases, patients with PMN undergo spontaneous remission with conservative approaches. Corticosteroids, alkylating agents and calcineurin inhibitors are recommended treatment options in persistent disease activity despite supportive therapies. Nevertheless, patients with refractory disease constitute an important clinical aspect of PMN, and uncontrolled proteinuria may culminate in rapid progression to end-stage renal disease. In recent years, several studies demonstrated the efficacy of rituximab as a treatment option in patients with refractory PMN; however, data regarding daily clinical practice of this agent is still needed. Therefore, we conducted a study using our registry data to evaluate the efficacy and safety of rituximab in patients with refractory PMN.

ELIGIBILITY:
Inclusion Criteria:

* Having biopsy-proven primary membranous nephropathy.
* Showing resistance to at least one set of prior therapies including corticosteroids, alkylating agents or calcineurin inhibitors.
* Having a history of rituximab use (375 mg/m2/wk for 2-4 weeks) following resistance aforementioned agents.

Exclusion Criteria:

* Not providing or withdrawing consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with primary membranous nephropathy who were treated using rituximab following resistance to at least one set of prior therapies including corticosteroids, alkylating agents or calcineurin inhibitors.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Complete Remission | 6 months
  Proteinuria <0.3 g/day, confirmed by two values at least 1 week apart, accompanied by a normal serum albumin concentration, and a normal serum creatinine.
Partial Remission | 6 months
  Proteinuria <3.5 g/day and a 50% or greater reduction from peak values, confirmed by two values at least 1 week apart, accompanied by an improvement or normalization of the serum albumin concentration and stable serum creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Halil Yazici, MD, Study Chair — Department of Internal Medicine, Istanbul Faculty of Medicine; Safak Mirioglu, MD, Principal Investigator — Department of Internal Medicine, Istanbul Faculty of Medicine
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dahan K, Debiec H, Plaisier E, Cachanado M, Rousseau A, Wakselman L, Michel PA, Mihout F, Dussol B, Matignon M, Mousson C, Simon T, Ronco P; GEMRITUX Study Group. Rituximab for Severe Membranous Nephropathy: A 6-Month Trial with Extended Follow-Up. J Am Soc Nephrol. 2017 Jan;28(1):348-358. doi: 10.1681/ASN.2016040449. Epub 2016 Jun 27. PMID 27352623